CLINICAL TRIAL: NCT06806215
Title: The Relationship Between Academic Burnout and Psychological Resilience Among Undergraduates Medical Students, Faculty of Medicine, Mansoura University
Brief Title: The Relationship Between Academic Burnout and Psychological Resilience
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: serial no: 0108323
Record Dates: First submitted 2025-01-26; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-05

CONDITIONS: Burnout; Resilience; Coping
Keywords: burnout; resilience; coping
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A cross sectional study of prevalence and correlates of burnout and resilience among indergraduate medical students

DETAILED DESCRIPTION:
A questionnaire based cross sectional study of The relationship between academic burnout and psychological resilience among undergraduates medical students, Faculty of Medicine, Mansoura University

ELIGIBILITY:
Inclusion Criteria:

- undergarduate medical students at Mansoura Faculty of Medicine

Exclusion Criteria:

* graduate students and interns

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: undergarduate medical students at Mansoura Faculty of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
burnout ,resilience | six months
  prevalence of burnout and resilience among undergraduate medical students

CONTACTS AND LOCATIONS:
Overall Officials: soha Rashed, Study Director — University of Alexandria
Locations (1):
- Faculty of Medicine Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
confidentiality